CLINICAL TRIAL: NCT05147909
Title: Impact of Dietary Phosphate Excess on Exercise Capacity and Visceral Adiposity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Wanpen Vongpatanasin, Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: STU-2021-1068
Record Dates: First submitted 2021-11-23; First posted 2021-12-07 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Physical Inactivity; Phosphate Overload; Visceral Obesity
MeSH Terms: conditions — Sedentary Behavior; Obesity, Abdominal | interventions — sodium phosphate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Investigational drug service at UT Southwestern will dispense Sodium Phosphate vs. NaCl tablets and the study subjects will be blinded to the type of supplement they receive.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sodium Phosphate (NaPO4) then sodium chloride (NaCl) (Experimental): Participants will be asked to take 2 capsules daily of Sodium Phosphate (containing a total of 500 mg of Pi, 372mg of sodium) ) for 4 weeks during the high Pi phase (total Pi intake 1,200 mg/d). Then, participants will be asked to take 2 capsules of Sodium Chloride (NaCl, containing a total of 372mg of sodium) to match Na content to Sodium Phosphate without extra Pi daily for 4 weeks during the low Pi phase (total Pi intake = 700 mg/d).
  Interventions: Dietary Supplement: Sodium Phosphate; Dietary Supplement: Sodium Chloride
- NaCl then NaPO4 (Experimental): Participants will be asked to take 2 capsules daily of Sodium Chloride (NaCl, containing a total of 372mg of sodium) for 4 weeks during the low Pi phase (total Pi intake = 700 mg/d). Then, participants will be asked to take 2 capsules of Sodium Phosphate daily for 4 weeks Sodium Phosphate (containing a total of 500 mg of Pi, 372mg of sodium) for 4 weeks during the high Pi phase (total Pi intake 1,200 mg/d).
  Interventions: Dietary Supplement: Sodium Phosphate; Dietary Supplement: Sodium Chloride

INTERVENTIONS:
Dietary Supplement: Sodium Phosphate — Sodium Phosphate 2 capsules daily (containing a total of 500 mg of Pi, 372mg of sodium)
  Other Names: NaPO4
Dietary Supplement: Sodium Chloride — Sodium Chloride 2 capsules daily (NaCl, containing a total of 372mg of sodium)
  Other Names: NaCl

SUMMARY:
Studies in mice demonstrated that dietary phosphate (Pi) loading that mimic the level of US adult consumption leads to reduced spontaneous locomotor activity, exercise capacity, and reduced resting metabolic rate when in normal mice by impairing skeletal muscle mitochondrial function and fat oxidation. However, relevance of this findings in humans remains unknown.

DETAILED DESCRIPTION:
The investigators will perform a randomized, crossover study to determine if lowering dietary Pi intake from 1,200 mg/day to recommended daily allowance (RDA) of 700 mg/day increases skeletal muscle ATP synthesis, raises exercise oxygen uptake (VO2) during cardiopulmonary testing. To ensure stable Pi intake prior to randomization, Pi consumption will be estimated by food recall during a run-in and washout phase for 2 consecutive days, using the Automated Self-Administered 24-Hour (ASA24®) Dietary Assessment Tool (https://epi.grants.cancer.gov/asa24/). After the run-in period, all participants will be maintained on a low Pi diet (700 mg/d) and a normal Na diet of approximately 3,128 mg/d throughout the study for 8 weeks. Subjects will also be randomized to receive Sodium Phosphate 2 capsules daily (containing a total of 500 mg of Pi, 372mg of sodium) for 4 weeks during the high Pi phase (total Pi intake 1,200 mg/d) vs 2 capsules of Sodium Chloride (NaCl, containing a total of 372mg of sodium) to match Na content to Sodium Phosphate without extra Pi daily for 4 weeks during the low Pi phase (total Pi intake = 700 mg/d). The total Na intake during the entire study will be at usual US consumption level of 3,500 mg/d. Investigational drug service at UT Southwestern will dispense Sodium Phosphate vs. NaCl tablets and the study subjects will be blinded to the type of supplement they receive.

During the periods of high and low Pi phases, the investigators will monitor 24-hr urinary Pi excretion (UPiV) to ensure adherence. Since approximately 70% of ingested Pi is absorbed and excreted in the urine, we expect 24-hr UPiV excretion to be approximately 840 mg during the high Pi phase and 490 mg during the low Pi phase. If 24-hr UPiV is < 800 mg during the high Pi diet or > 500 mg during the low Pi diet, the research dietitian will provide additional counseling to improve adherence to the menu plan. If needed, the research diet will be altered to be more compatible with the participant's preference.

24-hr urinary Pi, Na, K, Cr, and Ca excretion will be assessed after weeks 2 and 4 of the low and high Pi phases. Serum electrolytes and Pi will be monitored every 2 weeks. Serum FGF23, and soluble Klotho levels and cardiopulmonary testing and P31 MRS of quadriceps muscle will be obtained after 4 weeks on the study diet. The order of study supplement will be randomized. Subsequently, participants will stop the first study supplement and undergo washout for 2 weeks. After 2 weeks of washout, they will receive the 2nd study supplement. Measurement of skeletal muscle ATP synthesis and VO2 at rest and during exercise will be repeated in the same fashion.

ELIGIBILITY:
Inclusion Criteria:

The randomized crossover trial will be performed in on otherwise healthy subjects without diabetes mellitus, chronic kidney disease (CKD), preexisting cardiovascular disease or treatment with any vasoactive agent that might alter cardiovascular responses to exercise.

Exclusion Criteria:

1. history of cardiopulmonary disease or chronic kidney disease,
2. treatment with antihypertensive medications,
3. estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73m2, (4) diabetes mellitus or other systemic illness,

(5) pregnancy, (6) hypersensitivity to sodium phosphate, (7) any history of substance abuse or current cigarette use, (8) any history of psychiatric illness, (9) history of active malignancy, (10) serum phosphorus < 2.4 or > 4.5 mg/dL.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2022-09-14 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
oxygen uptake (VO2) during peak exercise | 4 weeks
  VO2 (ml of oxygen consumed /min) will be measured using a metabolic cart (Medgraphics) during exercise in a stationary bicycle. Standard breath-by-breath respiratory gases (VO2) will be measured at rest and after 3 minutes of steady state exercise at both 20 and 40 Watts using a cycle ergometer (Lode). Then, the partcipants will be asked to perform exercise to maximal level to obtain peak VO2.

SECONDARY OUTCOMES:
Resting ATP synthesis | 4 weeks
  Resting ATP synthesis (mM/min) will be measured using a magnetic resonance spectroscopy (MRS). The rate of exchange of high energy phosphates between phosphocreatine and ATP will be used to calculate resting ATP synthesis.
Phosphocreatine (PCr) depletion | 4 weeks
  PCr depletion (%) will be measured in the calf muscle after measurements of resting ATP synthesis by MRS. Participants will be asked to perform plantar flexion exercise for 1 min of foot-pushing against a magnet-compatible pulley system mounted on the scanner table constant workload (20% of estimated lean body weight at 2 s/cycle, 1 second of contraction/1 second of relaxation). Two bouts of exercise are performed by each subject with 10 min recovery between each bout and the results are averaged.
submaximal VO2 | 4 weeks
  VO2 (ml of oxygen consumed /min) will be measured using a metabolic cart (Medgraphics) during exercise in a stationary bicycle. Standard breath-by-breath respiratory gases (VO2) will be measured at rest and after 3 minutes of steady state exercise at both 20 and 40 Watts using a cycle ergometer (Lode) to obtain levels of sub maximal oxygen uptake
Cardiac output (CO) | 4 weeks
  CO (ml/min) will be measured at rest and during the same stationary bicycle exercise while VO2 is monitored, using an inert gas rebreathing method. The Innocor rebreathing system (Innovision A/S, Odense, Denmark) uses a combination of both an inert soluble gas (0.5% nitrous oxide) and an inert insoluble gas (0.1% sulfur hexafluoride) and has been shown to provide a reliable assessment of lung volumes and cardiac output non-invasively.

CONTACTS AND LOCATIONS:
Overall Officials: Wanpen Vongpatanasin, MD, Principal Investigator — Wanpen.Vongpatanasin@UTSouthwestern.edu
Locations (1):
- University of Texas Southwestern, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share de-identified data upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: 12 months after study is published